CLINICAL TRIAL: NCT07294040
Title: A Prospective Observational Study to Determine the Incidence and Risk Factors of Post-Induction Hypotension in Geriatric Oncologic Patients Undergoing General Anesthesia at a Tertiary Oncology Center
Brief Title: Incidence and Risk Factors of Post-Induction Hypotension in Geriatric Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Dolunay ARIK (Other)
Responsible Party: Sponsor-Investigator, Dolunay ARIK, Resident doctor, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Organization: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Other Study IDs: 2025-05/70
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-05

CONDITIONS: Post-induction Hypotension (PIH); Geriatric Patient; Oncologic Disease; Hemodynamic Effects of General Anesthesia; Risk Factors Associated With Anesthesia-Induced Hypotension
Keywords: Post-induction Hypotension; Perfusion Index (PI); Pleth Variability Index (PVI); geriatric patient; Oncologic Patients; General Anesthesia; Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Geriatric Oncologic Patients Monitored for Post-Induction Blood Pressure: This cohort includes geriatric patients (≥65 years) with a confirmed cancer diagnosis who are scheduled for surgery under general anesthesia. The focus of the study is on monitoring and evaluating post-induction blood pressure changes. Standard non-invasive monitoring (ECG, NIBP, SpO₂) will be applied, and blood pressure will be measured at predefined intervals in the first 20 minutes following anesthesia induction. The study aims to assess the frequency and determinants of post-induction hypotension in this patient population.

SUMMARY:
This observational clinical study aims to investigate the incidence and risk factors of post-induction hypotension (PIH) in geriatric cancer patients undergoing surgery under general anesthesia. PIH is defined as a drop in mean arterial pressure of ≥30% from baseline or below 65 mmHg within the first 20 minutes after anesthesia induction, prior to surgical stimulation.

The primary objective is to determine the frequency of PIH in elderly oncology patients. Secondary objectives include evaluating the association of PIH with age, ASA score, cancer type, oncological treatments (chemotherapy/radiotherapy), comorbidities, medication use, anemia, biochemical parameters, and preoperative perfusion index (PI) and pleth variability index (PVI).

Findings from this study are expected to contribute to improved perioperative management and to the development of tailored anesthesia protocols for geriatric oncology patients.

DETAILED DESCRIPTION:
This study will be conducted as a prospective observational trial at SBÜ Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Department of Anesthesiology and Reanimation, with the aim of evaluating the incidence and risk factors of post-induction hypotension (PIH) in geriatric oncology patients. The study will commence after institutional ethics committee approval, and written informed consent will be obtained from all participants.

Standard monitoring (ECG, non-invasive blood pressure, SpO₂) will be applied in the operating room. Pre-induction values will be recorded after a 5-minute rest period. Perfusion index (PI) and pleth variability index (PVI) will be measured using the Massimo Root® with Radical-7 monitor from the non-cannulated hand, with three consecutive readings averaged.

Demographic data (age, sex, height, weight, BMI), comorbidities, regular medications, type of malignancy, history of chemotherapy/radiotherapy, and preoperative laboratory values will be documented.

Anesthesia induction will be performed with propofol (1.5-2.5 mg/kg), fentanyl (1-2 μg/kg), lidocaine (1-1.5 mg/kg), and rocuronium (0.6 mg/kg). Maintenance will be achieved using sevoflurane (1.5-2%) or desflurane (5-6%), O₂/air mixture, and remifentanil (0.1-0.2 μg/kg/min). Drugs and doses used during induction will be recorded.

PIH is defined as hypotension occurring within the first 20 minutes after induction, prior to surgical stimulation. Criteria:

A ≥30% decrease in mean arterial pressure (MAP) compared to baseline or MAP < 65 mmHg Any interventions for hypotension (vasopressors, intravenous fluids) will be documented.

Blood pressure measurements will be obtained at six time points:

T0: Baseline, before induction T1: After induction, prior to intubation T2: 1 minute after intubation T3: 5 minutes after intubation T4: 10 minutes after intubation T5: 15 minutes after intubation

The study will be completed after the T5 measurement, covering the first ~20 minutes following anesthesia induction.

In this study, post-induction hypotension (PIH) will be defined as either a ≥30% decrease in mean arterial pressure (MAP) compared to the pre-induction baseline value, or MAP < 65 mmHg. The pre-induction MAP measured non-invasively will be taken as the baseline. During the first 20 minutes after induction (measured every 2 minutes), patients meeting either criterion will be classified into the "PIH present" group, while those without such changes will be classified as "PIH absent."

Sample size calculations were performed using G*Power 3.1:

For group comparisons: Assuming a medium effect size (Cohen's d = 0.5), 80% power, and α = 0.05, 64 patients per group (128 total) are required.

For categorical variables: With a medium effect size (Cohen's w = 0.3), 108 participants are required.

For logistic regression: Based on literature, the incidence of PIH was estimated at 20%. Assuming an Odds Ratio (OR) of 2.0, a two-tailed test with 80% power and α = 0.05 indicated that at least 113 participants are needed.

All statistical analyses will be conducted using SPSS or equivalent software, with a significance threshold of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥65 years of age

Patients with a diagnosis of cancer and scheduled for surgery

Ability and willingness to provide written informed consent

ASA physical status class II-IV

Exclusion Criteria:

Patients under 65 years of age

Patients without a confirmed oncologic diagnosis

Refusal to provide written informed consent

Patients undergoing regional anesthesia

Patients with tracheostomy or requiring multiple intubation attempts

History of peripheral arterial disease

Use of vasopressors before the start of surgery

Uncontrolled hypertension (blood pressure >180/110 mmHg)

Advanced heart failure (Ejection Fraction <40%)

Severe arrhythmias such as atrial fibrillation or significant ventricular arrhythmias that preclude reliable hemodynamic monitoring

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of geriatric patients (≥65 years) undergoing oncologic surgery at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Induction Hypotension (PIH) in Geriatric Oncologic Patients | From anesthesia induction to 15 minutes after intubation (≈ first 20 minutes post-induction)
  PIH defined as ≥30% decrease from pre-induction MAP or MAP < 65 mmHg at any measurement within the window (NIBP every 2 minutes). Outcome reported as the proportion of participants meeting PIH criteria.

SECONDARY OUTCOMES:
Association of Demographic, Oncologic, and Anesthetic Factors With Post-Induction Hypotension | From preoperative assessment to 20 minutes after anesthesia induction
  Secondary objectives include evaluating the relationship between PIH and patient characteristics such as age, ASA classification, cancer diagnosis, type of oncologic treatments received, comorbidities, regular medication use, preoperative anemia, selected biochemical parameters, perfusion index (PI) and pleth variability index (PVI) measurements, as well as the anesthetic induction method.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD publicly. Interested researchers may contact the principal investigator for data access

REFERENCES:
- [Background] Phillips AT, Deiner S, Mo Lin H, Andreopoulos E, Silverstein J, Levin MA. Propofol Use in the Elderly Population: Prevalence of Overdose and Association With 30-Day Mortality. Clin Ther. 2015 Dec 1;37(12):2676-85. doi: 10.1016/j.clinthera.2015.10.005. Epub 2015 Nov 6. PMID 26548320
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Background] Bloom MW, Hamo CE, Cardinale D, Ky B, Nohria A, Baer L, Skopicki H, Lenihan DJ, Gheorghiade M, Lyon AR, Butler J. Cancer Therapy-Related Cardiac Dysfunction and Heart Failure: Part 1: Definitions, Pathophysiology, Risk Factors, and Imaging. Circ Heart Fail. 2016 Jan;9(1):e002661. doi: 10.1161/CIRCHEARTFAILURE.115.002661. PMID 26747861
- [Background] Levin MA, Fischer GW, Lin HM, McCormick PJ, Krol M, Reich DL. Intraoperative arterial blood pressure lability is associated with improved 30 day survival. Br J Anaesth. 2015 Nov;115(5):716-26. doi: 10.1093/bja/aev293. Epub 2015 Sep 22. PMID 26395645
- [Background] Abebe MM, Arefayne NR, Temesgen MM, Admass BA. Incidence and predictive factors associated with hemodynamic instability among adult surgical patients in the post-anesthesia care unit, 2021: A prospective follow up study. Ann Med Surg (Lond). 2022 Jan 29;74:103321. doi: 10.1016/j.amsu.2022.103321. eCollection 2022 Feb. PMID 35145680